CLINICAL TRIAL: NCT05785689
Title: Autonomous Nervous System Regulated Anaesthesia: A Randomized Controlled Trial Comparing Dexmedetomidine and Placebo in Heart Rate Variability Monitored Children
Brief Title: Autonomous Nervous System Regulated Paediatric Anaesthesia With Dexmedetomidine or Placebo
Acronym: ANNA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense Patient Data Explorative Network (Other)
Responsible Party: Principal Investigator, Line Gry Larsen, Principal Investigator, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Eudract 202200094359
Record Dates: First submitted 2022-10-30; First posted 2023-03-27 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Postoperative Confusion; Postoperative Delirium; Postoperative Pain, Acute; Postoperative Complications
MeSH Terms: conditions — Emergence Delirium; Pain, Postoperative; Postoperative Complications | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DEX: Bolus dexmedetomidine 0,5 mcg/kg (Experimental): Intravenous infusion during first 10 minutes of anesthesia
  Interventions: Drug: Dexmedetomidine
- Placebo (PCB): Bolus isotonic saline (Placebo Comparator): Intravenous infusion during first 10 minutes of anesthesia
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — To reduce postoperative agitation
  Other Names: DEX
  Arms: DEX: Bolus dexmedetomidine 0,5 mcg/kg
Drug: Placebo — Placebo bolus saline
  Other Names: PCB
  Arms: Placebo (PCB): Bolus isotonic saline

SUMMARY:
The goal of this randomized, double blinded study is to examine in children whether postoperative agitation can be reduced.

The main question it aims to answer is Will optimized, monitor guided analgesic treatment and dexmedetomidine reduce postoperative agitation Participants will receive a standard anaesthesia regimen and on top of that, a titrable remifentanil infusion guided via Mdoloris Anastasia nociception index (ANI) monitor will be added. Additionally, the patients will receive either bolus placebo or bolus dexmedetomidine. The postoperative agitation measured via the Richmond agitation and sedation scale (RASS) score, will be compared. Secondary outcome measures including carbon dioxide trends will be made.

DETAILED DESCRIPTION:
Study protocol

Screening of eligible patients before procedure day All children assigned for evaluation for abdominal or urology procedures are primarily seen by surgeons in an ambulatory visit. This takes place in the months or weeks before surgery. If surgery for abdominal or urology issues is decided, the paediatric surgeons hand out a patient s folder about the present study. The patient information folder is seen in supplement 1. Line Gry Larsen (LGL) will attend the surgeon's ambulatory visits in the start-up phase, assisting the paediatric surgeons in what information to give by handing out patient information folders. It is not the intent that the paediatric surgeons should give the full information. If the parents/legal representative(s) consent to further contact, they sign a brief consent form for primary contact, including the preferred phone number and time frame, see supplement 2 The parents are then contacted by phone by one of the researchers within the assigned time frame, and the study is now introduced in full, in line with the information given in the patient information folder. There will be time for questions and careful consideration about participation. The researchers who provide the information to the families are all experienced within the field of anaesthesia, research, and Good Clinical Practice (GCP)-guidelines. If the parents show immediate interest in participating, the importance of bringing a signed power of attorney if one of the parents/legal representatives is not attending on the procedure day is emphasized.

Progress on procedure day

Information, consent, and randomization On the procedure day, one of the researchers again consults with the child and its parents/legal representatives in a private meeting room. They are offered the possibility to bring a bystander or be provided one. A summary of information about the study previously given by phone is done, including the right to withdraw consent. Questions are again encouraged. If the parents/legal representatives after receiving oral and written information agree on participation, consent forms are now signed and randomization is done to either placebo or intervention group, blinded for the participant, researcher, and other staff. The procedure is then performed that same day. Contact information is stored in the REDCap database for follow-up data, and to provide the family conclusions of the study after finalization.

Anaesthesia One or both parents or legal representatives follow the child to the operating theatre. Induction of anaesthesia is set as time = 0 and the first RASS score is registered. The child is then anaesthetized via inhalation of sevoflurane 8% on a mask while she or he is sitting with one of the parents. As soon as the child is asleep, the parents are shown to a waiting area. I.v access is obtained, and fentanyl 2-4 mcg i.v is given, and adjusted to fit the planned procedure. Airway management is typically done with a laryngeal mask aiming to keep the child spontaneous breathing throughout the procedure. Standard monitoring is applied: ECG, blood pressure cuff measuring, and fingertip oxygen saturation. Furthermore, all children are ANI monitored. A continuous infusion of remifentanil 0,5 mcg/kg/hour is started immediately and withheld for the entire procedure. Sevoflurane concentrations, airway pressure, and end-tidal carbon dioxide tensions, are noted. When all monitoring equipment is applied, a bolus infusion of the study drug (dexmedetomidine 0,5 mcg/kg or placebo) is given within the first 10 minutes. With ANI values < 50, a bolus of fentanyl of 1 mcg/kg or remifentanil 0,1 mcg/kg is given. Which drug is given, is assessed, and decided by the anaesthetist. The effect of this intervention is evaluated every five minutes and repeated if ANI is still < 50. Sevoflurane concentration is adjusted, guided by a clinical evaluation in a usual manner, guided by Minimum Alveolar Concentration (MAC) values 0,7-1,4. In the case of bradycardia or other arrhythmias, bolus dexmedetomidine (DEX) is immediately discontinued, and remifentanil (REMI) is withheld until baseline heart frequency is achieved. If longer-lasting bradycardia exists, iv. Atropine/kg bodyweight is given. To connect specific events to ANI values, the following are registered via the monitor: "infusions", "airway in", "incision", "bolus remifentanil", "bolus fentanyl", "neuraxial", "local anaesthesia", "bolus sevoflurane", "suture"," intense surgical stimuli"," bradycardia", "other [note in anaesthesia chart]", and "airway out".

All children receive standard premedication, consisting of oral or rectal diclofenac and paracetamol according to weight. Children will receive wound infiltration with local anaesthetics (bupivacaine 2.5 mg/mL) or a regional block while anaesthetized, when indicated.

The anaesthesia is terminated, the airway device is removed before leaving the operating theatre, and the child is then followed to the postoperative care unit (PACU). Even if project medication is withheld, data collected until that time and until discharged and follow-up, are included. In the case of an unexpected major change of standard procedure, e.g., a severe surgical complication resulting in surgeries far from normal procedures, ex. laparotomies, the patient will be excluded from the study.

The most time-critical point is on procedure day when general ward flow is to be balanced with appropriate time for the information, consent, randomization, and medicinal setup. The most time-critical data are the ANI values perioperatively and the importance of administering supplementary remifentanil boluses at the same time as when ANI values go below "50".

PACU stay Usual Face Legs Activity Cry Consolidation (FLACC) and Postoperative Nausea and Vomitation(PONV) scorings are done. For this study population, a supplementary RASS score is done every 15 minutes, a maximum nurse-Numeric Rating Scale (NRS)f, and a Paediatric Agitation and Emergence Delirium (PAED) score, each done once.

Follow up The parents/legal representatives will automatically receive a questionnaire via electronic mail as soon as the children are included in the study. In this, a "parent NRS", nausea, type, and dosage of pain killers are noted. If it is deemed too much of a task for the parent, the researchers can instead offer a follow-up phone interview and make the questionnaire orally with the parents. A questionnaire is seen in supplement 3. Due to the short half-life of the drugs used in this study, a long-term follow-up will not be done and participation in this study terminates at 24h.

Any protocol violations, adverse events (AEs), serious adverse events (SAEs), or suspected unexpected adverse reactions (SUSARS) are noted in a REDCap database and can be noted by all investigators. Additionally, SAE and SUSARS are noted in the SAE/SUSAR registration form as seen in supplement 4 The sponsor is notified of these automatically via an email notification provided by REDCap, or in case of breakdown, directly from the responsible researcher on procedure day. Common events such as challenges with obtaining i.v. access or laryngeal mask leak are not registered or stored in this study, as they are common and do have no correlation to study drugs or equipment.

Finally, the investigators wish to emphasize caution is taken, in creating a safe and comfortable atmosphere for both patients and their parents/legal representatives.

ELIGIBILITY:
Inclusion Criteria

* Children allocated for general anaesthesia in abdominal and urology setup.
* American Association of Anesthesiologists (ASA) score 1-2.
* Consent from both parents/legal representatives

Exclusion Criteria:

* ASA >2
* Missing consent from both parents/legal representatives.
* Known allergies or intolerances for remifentanil and dexmedetomidine.
* Intubation.
* Non fluently Danish speaking/reading parents/representatives

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Richmond Agitation Sedation Scale Score (RASS) | Once within the first minute at entering operating theatre
  Nurse evaluation of agitation/sedation on a scale from -5 (deeply sedated) to +4 (highly agitated)
Richmond Agitation Sedation Scale Score (RASS) | Once within the first minute at entering the postoperative care unit (PACU)
  Nurse evaluation of agitation/sedation on a scale from -5 (deeply sedated) to +4 (highly agitated)
Richmond Agitation Sedation Scale Score (RASS) | Every 15. minutes while admitted to postoperative care unit (PACU) and until discharge, within a time frame of maximum 240 minutes
  Nurse evaluation of agitation/sedation on a scale from -5 (deeply sedated) to +4 (highly agitated)

SECONDARY OUTCOMES:
Anaesthesia time consumption | From the minute of induction of anaesthesia minute of extubation, within a time phrame of 180 minutes
  Anaesthesia duration
Postoperative care unit (PACU) time consumption | From the minute of entering PACU area to the minute of discharge from hospital, within a time phrame of 400 minutes
  PACU duration
Total time consumption | From the minute of induction of anaesthesia to the minute discharge from hospital, within a time phame of 600 minutes
  Total admission duration
Total fentanyl dosage | From the minute of induction of anaesthesia to the minute discharge from hospital, within a time phame of 600 minutes
  Total dosage of fentanyl from whole hospital stay
total remifentanil dosage | From the minute of induction of anaesthesia to the minute discharge from hospital, within a time phame of 600 minutes
  Total dose remifentanyl infusion + boluses
Postoperative Nausea and vomiting (PONV) in Postoperative Care Unit (PACU) | From the minute of entering the PACU area to the minute of discharge from hospital, time phrame of maximum 400 minutes
  One maximum score within a 0 - 2 scale, "2" represents most PONV
Postoperative Nausea and vomiting (PONV) after discharge | From the minute of discharge from hospital until 24 hours after discharge from hospital. Time phrame of maximum 24 hours.
  One maximum score within a 0 - 2 scale during the first 24 hours after discharge. "2" represents most nausea.
Nurse - numeric Rating Score (nNRS) | From the minute of entering the PACU area to the minute of discharge from hospital, a time phrame of maximum 400 minutes
  Scale from 1-10 and "10" represents most pain. One maximum score for the entire postoperative care unit (PACU) stay
Parent - Numeric Rating Scale (pNRS) | From the minute of discharge from hospital until 24 hours after discharge from hospital. Time phrame of maximum 24 hours.
  Scale from 1-10, "10" is most pain. Maximum NRS estimated by parents
Face Leggs Agitation Cry Consolidation (FLACC) scale score | From the minute of entering the PACU area to the minute of discharge from hospital, a time phrame of maximum 400 minutes
  One maximum score, 0-10 points, 10 points represents most pain state
Paediatric Emergency Delirium Scale Score (PAED) scale score | From the minute of entering the PACU area to the minute of discharge from hospital, a time phrame of maximum 400 minutes
  One maximum score, 0-18 points, 18 points represents most delirium. Scoring done once during entire postoperative care unit (PACU) stay.
Paracetamol dosage | From admission to hospital until 24 hours after anesthesia, maximum of two days
  Total dose paracetamol given in relation to the anesthesia, both premedication and what is given from caretakers in hospital and parents the following day.
Voltaren dosage | From admission to hospital until 24 hours after anesthesia, time phrame of maximum of two days
  Total dose paracetamol given in relation to the anesthesia, both premedication and what is given from caretakers in hospital and parents the following day.
Other analgesics dosage | From admission to hospital until 24 hours after anesthesia, time phrame of maximum of two days
  Total dose of miscellaneous medications given in relation to the procedure/anesthesia
Propofol dosage | From the minute of induction of anaesthesia until care overtaken by postoperative care (PACU) nurses, within a time frame of 400 minutes
  Total dosage propofol given in relation to the anaesthesia
events | During anaeshtesia between induction and extubation, within a time frame of maximum 400 minutes
  Events during anesthesia: cough, movement, incision, extra fentanyl administration, bolus remifentanil, ANI < 50, suture, extubation, other
Carbondioxide tensions | Every five minutes during anaestesia, between induction and extubation, within a time phrame of maximum 400 minutes
  End-Tidal carbondioxide tension during anaeshtesia

CONTACTS AND LOCATIONS:
Overall Officials: Line G Larsen, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared to specific written requests to well defined elements and personal information about study participants will not be given.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 years
Access Criteria: Approved by principal investigator